CLINICAL TRIAL: NCT05956080
Title: Penicillin Allergy Delabeling Among Surgical Patients
Acronym: PenDel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 003
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Penicillin Allergy
MeSH Terms: interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allergy testing (Other)
  Interventions: Diagnostic Test: Allergy testing

INTERVENTIONS:
Diagnostic Test: Allergy testing — University Medicine Greifswald

SUMMARY:
Penicillin allergy testing among surgical patients

ELIGIBILITY:
Inclusion Criteria:

* surgical patients with reported penicillin allergy

Exclusion Criteria:

* missing consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Confirmed penicillin allergy | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Gibb, MD, Principal Investigator — University Medicine Greifswald; Christian S. Scheer, MD, Principal Investigator — University Medicine Greifswald

IPD SHARING:
Plan to Share IPD: Undecided